CLINICAL TRIAL: NCT06851832
Title: A Phase I/II Clinical Trial with Randomized, Blinded, Controlled Design to Evaluate the Safety and Immunogenicity of the Recombinant Herpes Zoster Vaccine (CHO Cell) in Healthy Populations Aged 40 Years and Older Post -vaccination
Brief Title: Clinical Trial of Recombinant Herpes Zoster Vaccine (CHO Cell) in Healthy Chinese Population Aged 40 Years and Older
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ab&B Bio-tech Co., Ltd.JS (Other)
Collaborators: Yither Biotechnology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VZV-ZHSW-01
Record Dates: First submitted 2025-02-25; First posted 2025-02-28 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Herpes Zoster; Herpes Zoster Vaccine
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Recombinant zoster Vaccine (CHO cell) (low adjuvant) (Experimental): It is used for vaccination of experimental vaccine group A subjects in phase I and II clinical trials
  Interventions: Biological: Recombinant zoster vaccine(CHO cell)(low adjuvant)
- Recombinant zoster Vaccine (CHO cell) (Experimental): It is used for vaccination of experimental vaccine group B subjects of phase I clinical trial , experimental vaccine group B1 and B2 subjects of phase II clinical trial
  Interventions: Biological: Recombinant Zoster Vaccine (CHO cell)
- Zoster Vaccine, Live (Active Comparator): It is used for vaccination of positive control group A1 and A2 subjects in phase Ⅱ clinical trial
  Interventions: Biological: Zoster Vaccine, Live
- Recombinant Zoster Vaccine (CHO cell) (Active Comparator): It is used for vaccination of positive control group B subjects in phase Ⅱ clinical trial
  Interventions: Biological: Recombinant Zoster Vaccine (CHO cell)
- Recombinant Zoster Vaccine (CHO cell) (Adjuvant control) (Placebo Comparator): It is used for vaccination of adjuvant control group subjects in phase Ⅰ clinical trial
  Interventions: Biological: Recombinant Zoster Vaccine (CHO cell) (Adjuvant control)
- normal saline (Placebo Comparator): Used in phase Ⅰ clinical trial; To maintain blinding, positive control group A1 and positive control group A2 received placebo on day 0 (for phase II clinical trial).
  Interventions: Biological: Normal Saline

INTERVENTIONS:
Biological: Recombinant zoster vaccine(CHO cell)(low adjuvant) — The dosage for each administration is 0.5 mL, containing 50 μg of gE, 0.25 mL of MF59, and 50 μg of CpG1018, administered intramuscularly into the deltoid muscle. A total of two doses will be given, with the second dose administered 30 days after the first dose.
  Arms: Recombinant zoster Vaccine (CHO cell) (low adjuvant)
Biological: Recombinant Zoster Vaccine (CHO cell) — The dosage for each administration is 0.5 mL, containing 50 μg of gE, 0.25 mL of MF59, and 100 μg of CpG1018, administered intramuscularly into the deltoid muscle.
  Vaccination Schedule 1: A total of two doses will be given, with the second dose administered 30 days after the first dose.
  Vaccination Schedule 2: A total of two doses will be given, with the second dose administered 60 days after the first dose [only applicable to the Phase II Experimental Vaccine Group B2].
  Arms: Recombinant zoster Vaccine (CHO cell)
Biological: Zoster Vaccine, Live — The dosage for each administration is 0.5 mL, containing not less than 4.3 lg PFU of varicella-zoster live virus, administered subcutaneously at the attachment site of the lower edge of the deltoid muscle on the outer side of the upper arm.
  A total of one dose will be given. To maintain blinding, the positive control group A1 will receive a placebo on Day 0 and the Zoster Vaccine, Live on Day 30. The positive control group A2 will receive a placebo on Day 0 and the Zoster Vaccine, Live on Day 60.
  Arms: Zoster Vaccine, Live
Biological: Recombinant Zoster Vaccine (CHO cell) — The dosage for each administration is 0.5 mL, containing 50 μg of gE and the AS01B adjuvant system [QS-21 (50 μg), MPL (50 μg), DOPC (1 mg), and cholesterol (0.25 mg)], administered intramuscularly into the deltoid muscle. A total of two doses will be given, with the second dose administered 60 days after the first dose.
  Arms: Recombinant Zoster Vaccine (CHO cell)
Biological: Recombinant Zoster Vaccine (CHO cell) (Adjuvant control) — The dosage for each administration is 0.5 mL, containing 0.25 mL of MF59 and 100 μg of CpG1018, administered intramuscularly into the deltoid muscle. A total of two doses will be given, with the second dose administered 30 days after the first dose.
  Arms: Recombinant Zoster Vaccine (CHO cell) (Adjuvant control)
Biological: Normal Saline — The dosage for each administration is 0.5 mL, containing 0.5 mL of NaCl solution, administered intramuscularly into the deltoid muscle. A total of two doses will be given, with the second dose administered 30 days after the first dose (applicable to Phase I clinical trial).
  To maintain blinding, subjects in the positive control A1 and positive control A2 groups will receive a placebo on Day 0 (applicable to Phase II clinical trial).
  Arms: normal saline

SUMMARY:
The objective of this study was to evaluate the safety, immunogenicity and immune persistence of recombinant herpes zoster vaccine (CHO cells) with different adjuvant doses in healthy people aged 40 years and older.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants aged 40 years or older at the time of enrollment.
* Voluntarily agrees to participate in the trial, fully understands, and signs the informed consent form.
* Able to attend all scheduled follow-ups and comply with the clinical trial protocol requirements to complete the trial.
* Female participants must meet the following criteria:1)Surgically sterilized or postmenopausal for ≥2 years, or women of childbearing potential (not menopausal or menopausal <2 years) with a negative pregnancy test and willing to use effective physical contraception (e.g., condoms, intrauterine device) from enrollment until 6 months after full immunization. 2)Agree not to breastfeed from enrollment until 6 months after full immunization.
* Axillary temperature ≤37.0°C.

Exclusion Criteria:

a Exclusion criteria for the first dose:

* A history of herpes zoster.
* A history of varicella or herpes zoster vaccination.
* Close contact with a varicella/herpes zoster patient within the past year.
* Received immunoglobulin and/or any blood products within 3 months before vaccination.
* Received immunosuppressive treatment within 3 months prior to vaccination (e.g., systemic corticosteroids for ≥14 days, at a dose ≥2 mg/kg/day or ≥20 mg/day of prednisone, or an equivalent dose of prednisone) (excluding inhaled, intra-articular, and topical steroids).
* A history of severe allergic reactions to any vaccine or medication (e.g., anaphylactic shock, allergic laryngeal edema, allergic purpura, thrombocytopenic purpura, local allergic necrosis reactions, severe urticaria, etc.), or a family history of severe allergies.
* Immunocompromised or diagnosed with congenital or acquired immune deficiency diseases, or infected with Human Immunodeficiency Virus (HIV).
* A history of seizures, epilepsy, encephalopathy (such as congenital brain malformation, brain trauma, brain tumors, cerebral hemorrhage, cerebral infarction [except for infarction without sequelae or lacunar infarction], brain infections, or brain damage caused by chemical drug poisoning), or psychiatric disorders, or a family history of psychiatric disorders; or other serious neurological diseases.
* Inadequate time interval between vaccination and other vaccines (e.g., inactivated or recombinant subunit vaccines within 14 days prior to vaccination, live attenuated vaccines, viral vector vaccines, or mRNA vaccines within 28 days prior to vaccination).
* Acute illness or an acute exacerbation of a chronic disease within 3 days prior to vaccination, or use of antipyretic, analgesic, or antihistamine medications within 3 days prior to vaccination.
* Suffering from severe infectious skin diseases.
* Ongoing or long-term alcohol and/or drug abuse history (Note: for the past three months, males drinking more than 14 standard drinks per week, females more than 7 standard drinks per week. One standard drink contains 14g of alcohol, equivalent to 360mL of beer, 45mL of liquor at 40% alcohol, or 150mL of wine. Drug abuse refers to the repeated or excessive use of drugs with dependence potential unrelated to recognized medical needs, for non-medical purposes).
* A history of thrombocytopenia or other coagulation disorders that may contraindicate intramuscular injection.
* Severe liver or kidney disease, complications from diabetes, severe cardiovascular diseases, or uncontrolled hypertension despite medication.
* Asplenia or functional asplenia, or any condition leading to splenectomy.
* Abnormal laboratory test results before the first dose, deemed clinically significant by the investigator (only applicable to Phase I).
* Currently participating in other experimental or unregistered clinical trials for products (drugs, vaccines, or devices), or planning to participate in another clinical trial before the end of this trial.
* A history of hematologic or lymphatic system diseases, such as unexplained lymphadenopathy or hematolymphatic lymphoma.
* A history of diagnosed potential immune-mediated diseases, autoimmune diseases, or Guillain-Barré syndrome.
* Any other condition deemed by the investigator to be unsuitable for participation in this clinical trial.

a Exclusion criteria for the second dose:

* Positive urine pregnancy test.
* Grade 4 adverse events related to vaccination.
* Severe allergic reactions occurring after vaccination.
* New findings or newly occurring conditions that meet the exclusion criteria after the first dose, with the investigator determining whether to terminate the trial vaccine administration.
* Other situations assessed by the investigator as requiring termination of vaccination.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 960 (Estimated)
Dates: Start 2025-02-16 (Actual); Primary Completion 2026-09-16 (Estimated); Study Completion 2028-09-16 (Estimated)

PRIMARY OUTCOMES:
The incidence of solicited local and systemic adverse events (AEs) within 0-14 days after each vaccine dose. | Within 14 days after each vaccine dose.
The incidence of unsolicited adverse events (AEs) within 0-30 days after each vaccine dose. | Within 30 days after each vaccine dose.
The incidence of laboratory abnormalities (including blood biochemistry, blood routine, urine routine and electrocardiogram) on Day 3 after each vaccine dose. | On Day 3 after each vaccine dose.（Applicable to Phase I only）
The incidence of serious adverse events (SAEs) and Adverse Events of Special Interest (AESI) from the vaccination of the first dose to 12 months after full immunization. | From the vaccination of the first dose to 12 months after full immunization.
The cell-mediated immune response rate of CD4+ T cells expressing at least two activation markers (IFN-γ, IL-2, TNF-α, CD40L) one month after full immunization. | One month after full immunization.（Applicable to Phase Ⅱ only）
  Detected using intracellular cytokine staining (ICS) by flow cytometry
The GMC/GMT, seroconversion rate, and GMI of anti-gE antibodies and anti-VZV antibodies one month after full immunization. | One month after full immunization.（Applicable to Phase Ⅱ only）
  Detected using enzyme-linked immunosorbent assay (ELISA).

SECONDARY OUTCOMES:
The GMC/GMT, seroconversion rate, and GMI of anti-gE antibodies and anti-VZV antibodies at 6, 12, 24, and 36 months after full immunization. | At 6, 12, 24, and 36 months after full immunization.（Applicable to Phase Ⅱ only）
  Detected using enzyme-linked immunosorbent assay (ELISA)
The cell-mediated immune response rate of CD4+ T cells expressing at least two activation markers (IFN-γ, IL-2, TNF-α, CD40L) before the second dose and at 6, 12, 24, and 36 months after full immunization. | Before the second dose and at 6, 12, 24, and 36 months after full immunization（Applicable to Phase Ⅱ only）
  Detected using intracellular cytokine staining (ICS) by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Zhiqiang Xie, Master, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Xiangcheng County Center for Disease Control and Prevention, Xuchang, Henan, China

IPD SHARING:
Plan to Share IPD: No